CLINICAL TRIAL: NCT04488809
Title: Comparison the Effects of Deep Water Running and Treadmill Running on Lower Extremity Anaerobic Exercise Performance in Sedentary Young Adults: A Randomized Controlled Study
Brief Title: Comparison the Effects of Deep Water Running and Treadmill Running
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Deniz Bayraktar, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DWRVSTR
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Sedentary Behavior
Keywords: Exercise; Running; Anaerobic Performance; Agility
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Water Running (Experimental): Participants in this group will perform running in a vertical position in water. The sessions will be held in deep pool where the feet of the participants will not touch the ground.
  Interventions: Other: Exercise
- Treadmill Running (Active Comparator): Participants in this group will perform running on a treadmill.
  Interventions: Other: Exercise
- Control (No Intervention): Participants in this group will not interfere regular exercise for 8 weeks.

INTERVENTIONS:
Other: Exercise — Exercise sessions will include 10 minutes of warming up, 30 minutes of loading, and 10 minutes of cooling down. The exercises will be performed two times in a week for eight weeks.
  Arms: Deep Water Running; Treadmill Running

SUMMARY:
The aim of this study is to compare the effectiveness of different exercise programs as 'Deep Water Running' and 'Treadmill Running' in sedentary young adults.

DETAILED DESCRIPTION:
Rapid and explosive movements such as jumping or stair climbing need anaerobic performance. Anaerobic performance is negatively affected by sedentary behaviour due to loss of muscle strength and endurance. Exercise is an effective method to increase muscle strength and physical performance.

Exercising in water has unique physiological characteristics such as buoyancy, hydrostatic pressure, and metacentric effect. In addition, exercising in high speeds in water leads strengthening. Deep water running is employed to imitate the running on land. It is advocated that deep water running might result additional benefits than running on land. Therefore, the effect of the present study is to compare the effectiveness of deep water running and treadmill running in sedentary young adults.

ELIGIBILITY:
Inclusion Criteria:

* Being sedentary according to International Physical Activity Questionnaire
* Consent of the participant

Exclusion Criteria:

* Problems related to musculoskeletal, neurologic, and cardiopulmonary systems in last six months
* Any contraindication to exercise in water (water fear, allergy to chlorine)
* No willingness to continue in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in lower extremity anaerobic performance | At baseline and 8 weeks later
  The lower extremity anaerobic performance will be measured by using Wingate Anaerobic Capacity Test. The average power (watt, watt/kg), and peak power (watt/watt/kg) will be recorded.

SECONDARY OUTCOMES:
Change in lower extremity strength | At baseline and 8 weeks later
  The strengths of M. Quadriceps Femoris, M. Gluteus Maximus, and M. Gastrocnemius will be assessed by using a hand-held dynamometer. Muscle strength will be recorded in kilograms.
Change in agility | At baseline and 8 weeks later
  T agility test will be used for evaluating agility. The time will be recorded for completing the test.
Change in trunk muscle endurance | At baseline and 8 weeks later
  Side bridge position will be employed to measure the trunk muscles endurance. The time until the failure in the position will be recorded.
Change in fatigue | At baseline and 8 weeks later
  Fatigue will be assessed by using Fatigue Severity Scale. It includes nine items, and each item is scored between 1-7 (1: totally disagree, 7: totally agree). Higher scores indicate higher levels of fatigue.
Change in total body mass | At baseline and 8 weeks later
  Total body mass will be measured by using bioelectrical impedance analysis and will be recorded in kilograms.
Change in fat mass | At baseline and 8 weeks later
  Fat mass will be measured by using bioelectrical impedance analysis and will be recorded in kilograms.
Change in fat free muscle mass | At baseline and 8 weeks later
  Fat free muscle mass will be measured by using bioelectrical impedance analysis and will be recorded in kilograms.
Change in basal metabolism rate | At baseline and 8 weeks later
  Basal metabolism will be measured by analyzing gas exchange in rest position. Oxygen consumption and carbon dioxide production will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Bayraktar, PT, PhD, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly BT, Roskin LA, Kirkendall DT, Speer KP. Shoulder muscle activation during aquatic and dry land exercises in nonimpaired subjects. J Orthop Sports Phys Ther. 2000 Apr;30(4):204-10. doi: 10.2519/jospt.2000.30.4.204. PMID 10778797
- [Background] Reichert T, Kanitz AC, Delevatti RS, Bagatini NC, Barroso BM, Kruel LF. Continuous and interval training programs using deep water running improves functional fitness and blood pressure in the older adults. Age (Dordr). 2016 Feb;38(1):20. doi: 10.1007/s11357-016-9882-5. Epub 2016 Feb 3. PMID 26841888
- [Background] Cuesta-Vargas AI, Buchan J, Arroyo-Morales M. A multimodal physiotherapy programme plus deep water running for improving cancer-related fatigue and quality of life in breast cancer survivors. Eur J Cancer Care (Engl). 2014 Jan;23(1):15-21. doi: 10.1111/ecc.12114. Epub 2013 Aug 16. PMID 23947581
- [Background] Cuesta-Vargas AI, Adams N, Salazar JA, Belles A, Hazanas S, Arroyo-Morales M. Deep water running and general practice in primary care for non-specific low back pain versus general practice alone: randomized controlled trial. Clin Rheumatol. 2012 Jul;31(7):1073-8. doi: 10.1007/s10067-012-1977-5. Epub 2012 Mar 29. PMID 22453844
- [Background] Wilber RL, Moffatt RJ, Scott BE, Lee DT, Cucuzzo NA. Influence of water run training on the maintenance of aerobic performance. Med Sci Sports Exerc. 1996 Aug;28(8):1056-62. doi: 10.1097/00005768-199608000-00017. PMID 8871917
- [Background] Broman G, Quintana M, Lindberg T, Jansson E, Kaijser L. High intensity deep water training can improve aerobic power in elderly women. Eur J Appl Physiol. 2006 Sep;98(2):117-23. doi: 10.1007/s00421-006-0237-2. Epub 2006 Aug 22. PMID 16924529
- [Background] Bayraktar D, Savci S, Altug-Gucenmez O, Manci E, Makay B, Ilcin N, Unsal E. The effects of 8-week water-running program on exercise capacity in children with juvenile idiopathic arthritis: a controlled trial. Rheumatol Int. 2019 Jan;39(1):59-65. doi: 10.1007/s00296-018-4209-8. Epub 2018 Nov 14. PMID 30430201
- [Background] Bar-Or O. The Wingate anaerobic test. An update on methodology, reliability and validity. Sports Med. 1987 Nov-Dec;4(6):381-94. doi: 10.2165/00007256-198704060-00001. No abstract available. PMID 3324256
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] Raya MA, Gailey RS, Gaunaurd IA, Jayne DM, Campbell SM, Gagne E, Manrique PG, Muller DG, Tucker C. Comparison of three agility tests with male servicemembers: Edgren Side Step Test, T-Test, and Illinois Agility Test. J Rehabil Res Dev. 2013;50(7):951-60. doi: 10.1682/JRRD.2012.05.0096. PMID 24301432
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Jebb SA, Cole TJ, Doman D, Murgatroyd PR, Prentice AM. Evaluation of the novel Tanita body-fat analyser to measure body composition by comparison with a four-compartment model. Br J Nutr. 2000 Feb;83(2):115-22. doi: 10.1017/s0007114500000155. PMID 10743490
- [Background] Vandarakis D, Salacinski AJ, Broeder CE. A comparison of COSMED metabolic systems for the determination of resting metabolic rate. Res Sports Med. 2013;21(2):187-94. doi: 10.1080/15438627.2012.757226. PMID 23541105